CLINICAL TRIAL: NCT06436261
Title: A Randomized, Multi-Center, Double-Blinded, Split-Face, Controlled Study Evaluating Procedure Pairing of a Post-Procedure Cream Versus a Comparator in Patients Treated With a Hybrid-Factional Laser for Facial Rejuvenation
Brief Title: Evaluating Procedure Pairing of a Post-Procedure Cream Versus a Comparator in Patients Treated With a Hybrid-Fractional Laser for Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RS-2021-03
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Photoaging; Wrinkle; Skin Laxity
Keywords: Post-Procedure; Hybrid Fractional Laser
MeSH Terms: conditions — Cutis Laxa | interventions — Sunscreening Agents; Sun Protection Factor

STUDY DESIGN:
Intervention Model Description: Randomized, Multi-Center, Double-Blinded, Split-Face, Controlled
Who Masked: Participant, Investigator
Masking Description: Subjects were randomly assigned to use the active post-procedure cream on one side of the face and the comparator moisturizer on the opposite side of the face.
  The products were packaged in the same container and labelled post-procedure cream. This was a double-blinded study, where the investigator, study subject, and other study personnel involved in the evaluation of efficacy or safety were blinded to the group during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Split-Face Application of Active (Experimental): Active (Experimental) Post-Procedure Cream
  Dosage Form: reverse emulsion (water in oil) cream containing bioactive ingredients, botanical actives, peptides, and antioxidants.
  Frequency of Dosage: Three times daily (morning, afternoon, and evening). Subjects were asked to apply to the face, forehead, under eyes, cheeks, upper lips, chin, and nose. The product was labelled with Right or Left depending on split-face randomization.
  Study Duration: 14 days. Active Post-Procedure Cream duration 14 days.
  Interventions: Procedure: Hybrid Fractional Laser; Other: Facial Cleanser; Other: Facial Moisturizer; Other: Sunscreen
- Split-Face Application of Comparator (Active Comparator): COMPARATOR:
  Dosage Form: moisturizer formulation
  Comparator Moisturizer Frequency of Dosage: Three times daily (morning, afternoon, and evening). Subjects were asked to apply to the face, forehead, under eyes, cheeks, upper lips, chin, and nose. The product was labelled with Right or Left depending on split-face randomization.
  Study Duration: 14 days. Comparator duration 14 days.
  Interventions: Procedure: Hybrid Fractional Laser; Other: Facial Cleanser; Other: Facial Moisturizer; Other: Sunscreen

INTERVENTIONS:
Procedure: Hybrid Fractional Laser — A hybrid fractional HALO™ laser treatment was performed after a 7-day washout period. Subjects were numbed for 30 minutes to 1 hour prior to the procedure with a topical numbing cream containing benzocaine, lidocaine, and/or tetracaine. After numbing was completed, patients received one full-face HALO™ laser treatment with settings 350/20/20.
  Other Names: HALO™ laser treatment
Other: Facial Cleanser — Subjects were to use the provided cleanser twice daily (morning and evening) during the 7-day washout period and 7-day post-procedure timeline.
  Other Names: Gentle Cleansing Lotion, Revision Skincare
Other: Facial Moisturizer — Subjects were to use the provided bland facial moisturizer as follows:
  WASHOUT PERIOD (7 days): After cleansing, 1-2 pumps were to be applied twice daily (morning and evening) to the full face avoiding the eye area
  POST-PROCEDURE (7 days): After applying the Post-Procedure Cream and Active Comparator based on split-face randomization, the facial moisturizer was to be applied twice daily (morning and afternoon).
Other: Sunscreen — During the 7-day washout period and 7-day post-procedure timeline, subjects were to apply the provided basic sunscreen in the morning and afternoon after applying facial moisturizer. Sunscreen was to be reapplied as needed throughout the day per FDA recommendations.
  Other Names: Aveeno Positively Mineral Sensitive Skin with sun protection factor (SPF) 40+

SUMMARY:
This randomized, multi-center, double-blinded, split-face, controlled clinical trial was conducted to investigate the tolerability, safety, and efficacy of a post-procedure cream when used immediately after hybrid-fractional laser treatment and for 7 days post-procedure with three times daily application in healthy female subjects aged 35-65 years with moderate to severe global face photodamage (score of 4 to 7 out of the 10-point Modified Griffiths' scale). Furthermore, this clinical trial compared the active post-procedure cream to a comparator moisturizer often paired with skin rejuvenation procedures. This is a cosmetic study with an FDA-regulated device.

A total of 16 healthy female subjects completed the study (8 subjects at both sites).

DETAILED DESCRIPTION:
This randomized, multi-center, double-blinded, split-face, controlled clinical trial was conducted to investigate the tolerability, safety, and efficacy of a post-procedure cream when used immediately after hybrid-fractional laser treatment and for 7 days post-procedure with three times daily application in healthy female subjects aged 35-65 years with moderate to severe global face photodamage (score of 4 to 7 out of the 10-point modified Griffith's scale). The ability of the post-procedure cream to soothe skin and improve patient downtime post-procedure was investigated by evaluating tolerability parameters (erythema, edema, dryness, burning, itching, stinging) over the course of the study. Furthermore, this clinical trial compared the active post-procedure cream to a comparator moisturizer often paired with skin rejuvenation procedures.

A 7-day washout period was required of all subjects prior to hybrid-fractional laser treatment. Tolerability (investigator: erythema, edema, dryness; subject: burning, itching, stinging) and safety were assessed through grading at screening, pre-procedure, post-procedure, post-procedure/post-product application, and days 1, 3, 5, and 7 post-procedure.

In addition, efficacy evaluation using the Modified Griffiths' scale was performed at screening, pre-procedure, and day 7 post-procedure. Self-assessment questionnaires were completed by subjects post-procedure/post-product application and days 1, 5, and 7 post-procedure. Clinical photography was completed at screening, pre-procedure, post-procedure/post-product application, and days 1, 3, 5, and 7 post-procedure.

A total of 16 healthy female subjects completed the study (8 subjects at both sites).

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects 35-65 years of age
* Fitzpatrick Skin Type I to III
* Moderate to severe global face photodamage (score of 4 to 7 out of the 10-point Modified Griffiths' scale, where 0 = none and 9 = severe)
* No known medical conditions that, in the Investigator's opinion, may interfere with study participation.
* Willing to discontinue all active topical facial products and only use the assigned test products for the duration of the study.
* Female subjects of childbearing potential must be willing to use a form of birth control during the study.

Exclusion Criteria:

* Nursing, pregnant, or planning a pregnancy during this study.
* Having undergone a chemical peel, dermabrasion, or microneedling (mechanical and radiofrequency) in the last 6 months; laser resurfacing (ablative, fractional, non-ablative) in the last 12 months
* Not willing to discontinue active topical facial products for 7 days prior to the Baseline Visit

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Investigator Tolerability | 7 days
  The primary tolerability endpoint will be Investigator Tolerability Assessment of erythema, edema, and dryness. A change in score of lack of significant change post-procedure/post-product application and days 1, 3, 5, and 7 post-procedure in comparison to immediately post-procedure indicates tolerability/safety of the test material.
  A four-point scale will be used with a lower score indicating a better outcome:
  0 = None
  1. = Mild
  2. = Moderate
  3. = Severe
Incidence of Adverse Events | 7 days
  The primary safety endpoint will be determined by the incidence and severity of adverse events in healthy subjects, including immediately post-procedure and throughout the length of the study.
Subject Tolerability | 7 days
  The subject tolerability endpoint will be Subject Tolerability Assessment of burning, itching, and stinging. A change in score of lack of significant change post-procedure/post-product application and days 1, 3, 5, and 7 post-procedure in comparison to immediately post-procedure indicates tolerability/safety of the test material.
  A four-point scale will be used with a lower score indicating a better outcome:
  0 = None
  1. = Mild
  2. = Moderate
  3. = Severe

SECONDARY OUTCOMES:
Self-Assessment Questionnaire | 7 days
  A change in response values at days 1, 5, and 7 compared to post-procedure/post-product application response values indicates an improvement. Baseline responses will be set to post-procedure/post-product application. Subjects are asked to rate statements based on a scoring system ranging from 5 (completely agree) to 1 (completely disagree). The best outcome is to Completely Agree with the statement / question being asked.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Burns, MD, Principal Investigator — Resurrect Skin MD; James Namnoum, MD, Principal Investigator — AYA™ Medical Spa
Locations (2):
- United States (2):
  - AYA™ Medical Spa, Atlanta, Georgia
  - Resurrect Skin MD, Dallas, Texas

REFERENCES:
- [Derived] Weir NM, Burns AJ, Kononov T, Zahr AS. A Novel Neurocosmetic Postprocedure Cream for Optimal Recovery and Tolerability From Energy-Based Devices. Lasers Surg Med. 2025 Dec;57(10):788-798. doi: 10.1002/lsm.70078. Epub 2025 Nov 24. PMID 41286587